CLINICAL TRIAL: NCT06298656
Title: Acute hemodynamiC Response To Carvedilol Predicts Survival in ACLF Patients - "ACT - C ACLF Study
Brief Title: Acute hemodynamiC Response To Carvedilol Predicts Survival in ACLF Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-ACLF-17
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Acute-On-Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — It is an observational study.

SUMMARY:
Clinically significant portal hypertension (CSPH) is defined as HVPG >10 mmHg. Patients with CSPH are at risk of developing esophageal varices and clinical decompensation (variceal bleeding, ascites, jaundice, encephalopathy), which mark the transition from compensated stage to a stage of the disease (decompensated) associated with higher mortality (1). HVPG is calculated by subtracting the free hepatic venous pressure (FHVP), a measure of systemic pressure, from the wedged hepatic venous pressure (WHVP), a measure of hepatic sinusoidal pressure. HVPG is surrogate marker in many clinical applications such as gold standard test to evaluate presence and severity of portal hypertension (PHT) diagnosis, risk stratification, monitoring of the patients on beta blockers (2). Non selective beta-blockers like propranolol and carvedilol are indicated in adults for primary and secondary prophylaxis of variceal hemorrhage. Acute hemodynamic response to intravenous propranolol with HVPG values coming down to <12 mm Hg or reduction to >20% from baseline have been shown to be associated with reduced long term risk of variceal bleed. Hence we are planning the current work to study the Acute hemodynamiC response To Carvedilol predicts survival in ACLF patients - "ACT - C ACLF study

DETAILED DESCRIPTION:
To assess whether Acute hemodynamic response to oral Carvedilol can predict short term outcome in ACLF patients.

• To determine the best cut off to define acute hemodynamic response in ACLF patients

Primary outcome - Predictive value of acute HVPG change by carvedilol for 28 day transplant free survival in patients of ACLF

Secondary outcome -

(1) Complications [PHT related bleed, AKI, infections, HE, Hypotension, Cardiac side effect] within 90 days (2) Transplant-free survival rate at 90 days (3) Correlation with evolution of AARC score by 2 week

(b) Methodology

Study population: Patients of age 18 to 70 years with ACLF fulfilling the conditions as per inclusion and exclusion criteria

Baseline parameters that will be recorded:

1. Baseline characteristics:
2. History and etiology of liver disease
3. Symptomatology, Evidence of decompensation (jaundice, encephalopathy, ascites, infections, variceal bleed etc)
4. Clinical and demographic profile
5. Endoscopy

Stopping rule of study:

1. Progression to exclusion criteria
2. In case of hypotension(<90/60mmHg) or Heart Rate <60 after carvedilol
3. Potential liver transplant within 90 days

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 yrs
2. ACLF diagnosis (AARC criteria)

Exclusion Criteria:

1. Contraindications to NSBB (Heart rate < 65 /min, BP < 110/65 mm Hg, Asthma, Heart failure, AKI, Large ascites, SBP, S. Na < 125meq/l)
2. PVT
3. HCC
4. BCS
5. HE grades 2-4
6. NSBB therapy within 5 days
7. Pregnancy
8. Lactation
9. Planned for LT in the next 12 weeks
10. No consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of age 18 to 70 years with ACLF fulfilling the conditions as per inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-10 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Predictive value of acute HVPG change by carvedilol for 28 day transplant free survival in patients of ACLF | 28 days

SECONDARY OUTCOMES:
Complications [PHT related bleed, AKI, infections, HE, Hypotension, Cardiac side effect] within 90 days | 90 days
Transplant-free survival rate at 90 days | 90 days
Correlation with evolution of AARC score by 2 week | 2 week

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided